CLINICAL TRIAL: NCT06728501
Title: Diabetes Education for Patients With Type 2 Diabetes in Turkmenistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Klaus Parhofer, Prof of Endocrinology and Metabolism, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiabetesEducationTurkmenistan
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes education (Active Comparator): Patients receive diabetes education
  Interventions: Behavioral: Diabetes education
- Control (No Intervention): Patients receive no diabetes education

INTERVENTIONS:
Behavioral: Diabetes education — Patients receive 5 hours of diabetes education
  Arms: Diabetes education

SUMMARY:
The aim of the study is to investigate whether structured diabetes mellitus education leads to improved blood glucose control in Turkmenistan.

DETAILED DESCRIPTION:
Diabetes education is not routinely carried out in Turkmenistan. The aim of the study is to investigate whether patients with type 2 diabetes benefit from an International Diabetes Federation (IDF) based education program. Patients will be randomized into a education group and a control group. The education group will receive 4 - 5 hours of education and the control group will only receive general information about diabetes mellitus. After 6 months, it is checked whether the change in the HbA1c value differs between the two groups. Additinal paremeters such as blood pressure, diabetes knowledge and lipids will also be evaluated (secondary parameters).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes

Exclusion Criteria:

* type 1 diabetes
* diabetes duration < 1 year
* severe comorbidities
* abuse of alcohol or drugs
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- International Center of Surgery and Endocrinology, Ashgabat, Turkmenistan, Ashgabat, Turkmenistan

IPD SHARING:
Plan to Share IPD: No